CLINICAL TRIAL: NCT02081768
Title: Assessment of the Efficacy of Stereotactic Intracavitary Instillation of 90yttrium Colloid for Treatment of Cystic Lesions of the Pituitary and Surrounding Areas (Sellar/Parasellar Region)
Brief Title: 90Yttrium Colloid for the Treatment of Cystic Sellar/Parasellar Tumors
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: David Clarke (Other)
Responsible Party: Sponsor-Investigator, David Clarke, Neurosurgeon, Nova Scotia Health Authority
Organization: Nova Scotia Health Authority (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Yttrium2014
Record Dates: First submitted 2014-03-05; First posted 2014-03-07 (Estimated); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Cystic Tumors of the Sellar/Parasellar Region
Keywords: Rathke's cleft cyst, pituitary cysts; cystic craniopharyngiomas
MeSH Terms: conditions — Central Nervous System Cysts

STUDY DESIGN:
Intervention Model Description: 90Yttrium colloid
Masking Description: Open label
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 90yttrium colloid (Experimental): 90 Yttrium colloid will be inserted into the cystic cavity. Based on clinical expertise, the treating neurosurgeon will determine the appropriate surgical procedure for each patient on an individual basis which will be reflected in the surgical consent the patient is presented and signs.
  Interventions: Radiation: 90yttrium colloid

INTERVENTIONS:
Radiation: 90yttrium colloid — 90yttrium colloid will be inserted into a sellar/parasellar cyst

SUMMARY:
There is no consensus in the literature on the best way to treat cystic lesions of the pituitary area. Patients who are symptomatic from these tumours are rare. The cystic form of tumours present special challenges since traditional treatment modalities (surgery and/or external radiation) are often not able to completely remove or treat the cyst wall without major morbidity or even mortality.

There is no 'best practice' for the treatment of cystic tumours per se. Treatments available to patients with cystic sellar/parasellar tumours include conservative management using a 'wait and scan' approach, cyst drainage, and cyst removal via transsphenoidal and/or craniotomy approach (i.e. open surgery). Over the last 10 years we have treated approximately 8 patients with intracystic radiotherapy. All of these patients continue to be monitored clinically and radiologically and all have done well with stable regression of the cysts and no new neurological deficits. Over the past 2 years, 90yttrium colloid has been provided to CDHA through Health Canada's Special Access Program (SAP). It has only been of recent that Health Canada has requested a clinical trial to assess the benefit of intracystic radiotherapy over other available treatment options.

The experimental treatment being proposed is the stereotactic intracavitary instillation of 90yttrium colloid for treatment of cystic lesions of the pituitary (sellar) and surrounding areas (parasellar).

DETAILED DESCRIPTION:
Surgical procedures will be performed as standard of care. The treating neurosurgeon (Dr. David B. Clarke) will determine surgical parameters based on his clinical expertise.

ELIGIBILITY:
Criteria

Ages Eligible for Study: 17 years of age or older Genders Eligible for Study: Both Accepts Healthy Volunteers: No

Inclusion Criteria

Patients who meet all of the following criteria are eligible for enrollment as study participants:

1. Patients 17 years of age or older.
2. Cystic sellar, suprasellar, parasellar or intrasellar masses diagnosed by histology, cytology or neuroimaging.
3. Tumour measurements and/or tumour volume can be calculated.
4. Patients who require surgical intervention as determined by the treating neurosurgeon.
5. Being a patient managed in the Halifax Neuropituitary Program surgical clinic.
6. Willingness to undergo surgery and give informed surgical consent.
7. Willingness to provide informed consent for study participation.

Exclusion Criteria

Patients who meet any of these criteria are not eligible for enrollment as study participants:

1. Neurosurgeon's assessment that surgical procedures hold unacceptable operative risk.
2. Having a solid tumour.
3. Pregnant or breast feeding at time of surgical consent and/or surgery.
4. Hypersensitivity, allergies or contraindication to the used radiopharmaceutical agent (90yttrium colloid).

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-06; Primary Completion 2031-06-30 (Estimated); Study Completion 2031-10-31 (Estimated)

PRIMARY OUTCOMES:
Cyst shrinkage | 12 months after treatment
  Decreased cyst volume on MRI + resolution of clinical symptoms

SECONDARY OUTCOMES:
Localization of intracystic 90yttrium colloid by PET-CT | Within 3 weeks of treatment
  Visualization of 90 yttrium colloid within the cyst

CONTACTS AND LOCATIONS:
Overall Officials: David Clarke, Principal Investigator — Capital District Health Auhtority
Locations (1):
- Halifax Infirmary, Halifax, Nova Scotia, Canada